CLINICAL TRIAL: NCT04418310
Title: Lay Open and Curettage Versus Endoscopic (E.P.Si.T) Method in the Treatment of Sacrococcygeal Pilonidal Sinus Disease
Brief Title: Intervetional Lay Open and Curettage Versus Endoscopic (E.P.Si.T) Method in the Treatment of Sacrococcygeal Pilonidal Sinus Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Epsit Pilonidal sinus
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-05

CONDITIONS: Endoscopic Pilonidal Sinus
MeSH Terms: interventions — Curettage; Endoscopy; Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lay open and curettage (Active Comparator): Lay open and curettage in Pilonidal sinus
  Interventions: Procedure: Lay open and curettage
- Endoscopic (E.P.Si.T) method (Active Comparator): Endoscopic (E.P.Si.T) method in the treatment of sacrococcygeal pilonidal sinus disease
  Interventions: Procedure: Endoscopic (E.P.Si.T) method

INTERVENTIONS:
Procedure: Lay open and curettage — Lay open and curettage
  Arms: Lay open and curettage
Procedure: Endoscopic (E.P.Si.T) method — Endoscopic (E.P.Si.T) method
  Arms: Endoscopic (E.P.Si.T) method

SUMMARY:
Aim of the work To compare lay open technique versus Endoscopic pilonidal sinus treatment as regards recurrence rate, operative data, postoperative pain, intra and postoperative complications, healing time and return to daily activity

DETAILED DESCRIPTION:
Introduction Pilonidal sinus is a very common inflammatory disease of gluteal region (McCallum et al., 2008). Its incidence is 26/100,000 and it usually occurs in working males of age 15 to 30.

The disease itself dates back to 1833 when Herbert Mayo, British Physiologist, Anatomist and Surgeon described it as a sinus containing hair follicles located in the sacrococcygeal region in a woman.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders with symptoms from sacrococcygeal pilonidal sinus were included in our study.

Exclusion Criteria:

* Abscess formation 2. Immunodeficiency. 3. Patients with congenital asymptomatic pits. 4. Patient with psychiatric disease disabling surgical intervention. 5. Pregnant females

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | one year
  recurrence rate of pilonidal sinus symptoms after healing

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt